CLINICAL TRIAL: NCT00672191
Title: A Phase II Study Testing the Activity and Safety of AGS-004 as an Immunotherapeutic in Successfully ART-Treated Subjects Infected With HIV-1 in Combination With ART Followed by ART Interruption
Brief Title: Phase II Study of AGS-004 as an Immunotherapeutic in Antiretroviral Therapy (ART)-Treated Subjects Infected With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-004-001
Record Dates: First submitted 2008-05-05; First posted 2008-05-06 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infections
Keywords: HIV; Human immunodeficiency virus; Immunodeficiency Virus, Human; HIV-1; ART; antiretroviral therapy; HAART; highly active retroviral therapy; cluster of differentiation CD 4+ T cell counts; HIV-1 Subjects successfully ART treated; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: AGS-004

INTERVENTIONS:
Biological: AGS-004 — HIV-1 Immune Therapy

SUMMARY:
The purpose of this study is to examine the ability of AGS-004 to control HIV-1 replication and to determine if HIV-1 immunotherapy made with dendritic cells is safe and well tolerated, to determine if immunotherapy increases the body's immune response to HIV-1; and, to determine if after stopping anti-HIV drugs, immunotherapy can control the HIV-1 virus.

DETAILED DESCRIPTION:
Although chronic ART raises cluster of differentiation CD 4+ T cell counts and improves immune function, the immune systems' ability to control HIV-1 replication is not improved. AGS-004 is an immunotherapeutic agent made from autologous DCs co electroporated with amplified in vitro transcribed (IVT) ribonucleic acid (RNA) encoding CD40L and with IVT RNA encoding three or four autologous HIV-1 antigens. The HIV-1 RNA is derived from the plasma sample taken immediately prior to the initiation of ART.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age
* HIV-1 infection
* Subjects must be on their first ART regimen for at least 3 months: 2 NRTIs together with an NNRTI and/or at least 1 PI (prior changes to ART regimen are allowed if due to tolerability, guideline change, or to simply dosing but not for viral control)
* Durable viral suppression (below limit of detection) for at least 3 months prior ot Screening
* CD4+ T cell count ≥ 450 cells/mm3 for at least 90 days immediately prior to Screening
* Availability of ≥ 1.2 mL of continually frozen plasma (may have been thawed and refrozen only once) drawn no more than 90 days before starting ART and preferably within 30 days.
* Pre-ART plasma HIV-1 RNA levels of ≥ 15,000 copies/mL at the time the plasma was archived before commencing ART
* Pre-ART nadir CD4+ T cell count ≥ 200 cells/mm3 (cell count of < 200 cells/mm3 on one occasion is allowed if subsequent pre-ART CD4+ cell counts were > 200 cells/mm3 on at least two time points.
* Laboratory values obtained at Screening and confirmed just prior to Baseline Day 1:

  * Creatinine ≤ 1.5 x upper limit of normal (ULN);
  * AST (SGOT), ALT (SG'PT), and alkaline phosphatase ≤ 3 x ULN;
  * ANC ≥ 750 cells/mm3;
  * Hemoglobin ≥ 10 g/dL; and,
  * Platelet count ≥ 75,000/mm3
* Female subjects of reproductive potential must have a negative serum or urine pregnancy test with a sensitivity of at most 50 mIU/mL performed within 30 days prior to Screening.
* All subjects must agree not to participate in a conception process and use contraception.
* Ability to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements.
* Voluntary informed consent given to participate in the study.
* Successful RNA amplification of at least 3 antigens (must include Gag).

Exclusion Criteria:

* HIV-2 antibody positive.
* Positive test for other infectious diseases including:

  * clinically active, untreated syphilis (positive rapid plasma regain test (RPR)
  * clinically active hepatitis B infection (positive Hep B surface antigen HBsAg)
  * active hepatitis C infection or any history of hepatitis C infection
  * positive test for HTLV Type I or Type II antibody
* Any acute infection or serious medical illness within 14 days prior to study entry
* History of lymph node irradiation or dissection
* Pregnancy or breast-feeding
* Previous use of any HIV-1 immunotherapy, including IL-2
* Use of hydroxyurea within 30 days prior to Screening
* Immunodeficiency other than HIV-1 or requirements to take immuno-modulating concomitant medications
* Known allergy or sensitivity to the investigational immunotherapy or its formulation
* Use of systemic corticosteroids and use of topical steroids over a total area exceeding 15 cm2 within 4 weeks of Screening or anticipated need for periodic use of corticosteroids during the study
* Receipt of any immune modulators or suppressors within 30 days of Screening
* Active autoimmune disease such as:

  * Rheumatoid arthritis
  * Inflammatory bowel disease
  * Systemic lupus erythematosis
  * Ankylosing spondylitis
  * Hashimoto's disease
  * Scleroderma
  * Multiple sclerosis
  * Autoimmune hemolytic anemia
  * Immune thrombocytopenic purpura
* Type I diabetes mellitus (insulin therapy for Type II diabetes is permitted)
* Participation in another clinical trial within 30 days of Screening or use of investigational agents (previous use of expanded access ARTs is permitted)
* Body weight less than 30 kg.
* Changes in ART regimen due to virologic failure (not including toxicities)
* Presence of factors predicting insufficient adherence to the protocol.
* Any condition that in the assessment of the investigator would indicate that it is not in the best interest of the subject or incompatible with the any aspect of the study design, treatment plan, and study objectives for a subject to participate.
* History or other evidence of severe illness, malignancy, or any other condition that would make the subject, in the opinion of the investigator, unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Ability of AGS-004 therapy to improve immune control of HIV-1 replication | Study Week 26 through end of study

SECONDARY OUTCOMES:
Change in plasma HIV-1 RNA set point | Study Week 26 through end of study
T cell responses to AGS-004 therapy and exploratory studies to investigate the mechanism of action of AGS-004. | Study Week 26 through end of study
Safety and tolerability of AGS-004 | Study Week 26 through end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Mona Loutfy, MD, Principal Investigator — Maple Leaf Clinic; Cecile Tremblay, MD, Principal Investigator — CHUM- Hotel Dieu de Montreal; John Gill, MD, Principal Investigator — Southern Alberta Clinic; Jean-Guy Baril, MD, Principal Investigator — Clinque Medical du Quartier Latin; Sylvie Vezina, MD, Principal Investigator — Clinque medicale l'Actuel; Jonathan B Angel, MD, Principal Investigator — The Ottawa Hospital; Sharon Walmsley, MD, Principal Investigator — UHN; Fiona Smaill, MD, Principal Investigator — Hamilton Health Sciences Corporation; Anita Rachlis, MD, Principal Investigator — Sunnybrook Health Sciences Center; Julio Montaner, MD, Principal Investigator — Providence Health Care Society; Jeffrey Jacobson, MD, Principal Investigator — Partnership Comprehensive Care Practice
Locations (12):
- Practice Comprehensive Care Practice Div of Onfectious Disease & HIV Med, Philadelphia, Pennsylvania, United States
- Canada (11):
  - Southern Alberta Clinic, Calgary, Alberta
  - Providence Health Care Society / The University of British Columbia / BC Centre for Excellence in HIV/AIDS, Vancouver, British Columbia
  - Hamilton Health Sciences - McMaster University Medical Centre, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Maple Leaf Clinic, Toronto, Ontario
  - UHN, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique Medical du Quartier Latin, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - CHUM, Montreal, Quebec